CLINICAL TRIAL: NCT02018666
Title: ZEPHYR: Multicenter, Prospective, Randomized, Open-label Study in Consecutive Patients Hospitalized for Acute Respiratory Failure Requiring Mechanical Ventilation With Endotracheal Tube. This Study Compared Two Ventilation Modes: NAVA Mode and Spontaneous Breathing With Inspiratory Pressure Support (the Latter is Considered as the Reference Ventilation Mode).
Brief Title: Study Comparing Two Ventilation Modes NAVA (Neurally Adjusted Ventilatory Assist) Mode and Spontaneous Breathing With Inspiratory Pressure Support (IPS) Mode in Consecutive Patients Hospitalized for Acute Respiratory Failure Requiring Mechanical Ventilation With Endotracheal Tube.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinact (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N° 2011-001; 2011-A00559-32 (Other: ANSM)
Record Dates: First submitted 2013-12-11; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Acute Respiratory Failure

ARMS (2):
- spontaneous NAVA mode (Experimental)
  Interventions: Device: NAVA endotracheal tube
- Inspiratory pressure support (IPS) (Active Comparator)
  Interventions: Device: NAVA endotracheal tube

INTERVENTIONS:
Device: NAVA endotracheal tube

SUMMARY:
This is a multicenter, prospective, randomized, open-label study which compared two ventilation modes: spontaneous NAVA mode and spontaneous breathing with IPS mode (the latter is considered as the reference ventilatory mode) in patients admitted to the ICU for acute respiratory failure and ventilated with an endotracheal tube. NAVA mode allows to minimize patient-ventilator disharmony with acceptable tolerance and to preserve spontaneous ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ventilated with endotracheal tube for more than 24 hours
* Return for at least 30 minutes to spontaneous ventilation allowing IPS with a level of pressure support <30 cm H2O;
* Level of sedation =< 4 on the Ramsay scale in the absence of medical decision to increase the level of sedation;
* Fraction of inspired oxygen (FiO 2) =< 50% with a positive end-expiratory pressure (PEEP) =< 8 cm H2O;
* Absence of administration of high-dose vasopressor therapy defined by:

  1. norepinephrine > 0.3 mcg / kg / min;
  2. dopamine > 10 mcg / kg / min;
* Estimated duration of mechanical ventilation > 48h00

Exclusion Criteria:

* Contraindication to the implementation of the NAVA endotracheal tube, ie any contraindication to the implementation of a gastric tube or to the repositioning of a tube already in place:

  1. Recent gastrointestinal suture ;
  2. Esophageal varices rupture with gastrointestinal bleeding within 4 days prior to inclusion;
* Therapeutic limitation or active treatment discontinuation;
* Pregnant women;
* Minors;
* Protected adults;
* Patient already included in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the benefit of NAVA mode as compared to IPS mode in terms of duration of spontaneous ventilation 48 hours after inclusion. | Continuous recording during 48 hours following the intubation
  The time spent in different modes of spontaneous ventilation (NAVA, IPS) and controlled ventilation (VAC controlled pressure) will be measured. The primary endpoint will be the proportion of patients remaining in spontaneous ventilation after the first 48 hours.

SECONDARY OUTCOMES:
Reduction of patient / ventilator disharmony, measured during the first 48 hours with the disharmony index | Continuous recording during the first 48 hours
Real-time spent in NAVA mode and frequency of returns in a controlled mode (controlled ventilation VAC). | Continuous recording during the first 48 hours
  Feasibility of the initiation of mechanical ventilation in NAVA mode and feasibility of prolonged mechanical ventilation in NAVA mode
Earnings on the "breathing comfort" | Continuous recording during the first 48 hours
Earnings on sleep architecture | Continuous recording during the first 48 hours
  Total sleep time; Number of arousals per hour; Duration of stage IV sleep ; Duration of Rapid Eye Movement (REM) sleep.
Tolerance | Continuous for the duration of ICU stay, an expected maximum of 14 days
  * Adverse events associated with the use of the device.
  * Incidence of ventilator-acquired pneumonia.
  * Duration of ICU stay.
  * Duration of hospital stay.
  * Mortality in the ICU.
  * Hospital mortality.

OTHER OUTCOMES:
Number of implementation failure of the NAVA endotracheal tube. | For each patient, the success or failure of the endotracheal tube implementation will be evaluated, this for the entire duration of the study estimated to 18 months
Number and duration of automatic switch into IPS mode | Continuous recording until extubation or D14 maximum
Number of Permanent discontinuation of NAVA ventilation mode | Continuous recording during the first 48 hours
Comfort of the device measured by a visual analog scale. | At the extubation or at D14 maximum
  Tolerance of the device
Side effects associated with the use of the system | Continuous for the duration of ICU stay, an expected maximum of 14 days
  Device movements Endotracheal tube obstruction Lesion of the oral or nasal mucosa

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Hopital L'Archet 1, Nice, Alpes Maritimes
  - Hopital de la CROIX ROUSSE, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon Sud, Lyon, Auvergne-Rhône-Alpes
  - Hopital PELLEGRIN, Bordeaux, Gironde
  - Groupe Hospitalier Sud - Hôpital Haut-Leveque - Maison du Haut-Leveque, Pessac, Gironde
  - Hôpital Dupuytren, Limoges, Haute Vienne
  - Hopital Saint-Eloi - CHU MONTPELLIER, Montpellier, Herault
  - Hopital Larrey- CHU D'ANGERS, Angers, Maine Et Loire
  - Hopital de la Cote de Nacre - CHU de CAEN, Caen, Normandy
  - Hopital d'Estaing, Clermont-Ferrand, Puy de Dome
  - Hôpital de la Pitié Salpetrière, Paris, Île-de-France Region

REFERENCES:
- [Derived] Demoule A, Clavel M, Rolland-Debord C, Perbet S, Terzi N, Kouatchet A, Wallet F, Roze H, Vargas F, Guerin C, Dellamonica J, Jaber S, Brochard L, Similowski T. Neurally adjusted ventilatory assist as an alternative to pressure support ventilation in adults: a French multicentre randomized trial. Intensive Care Med. 2016 Nov;42(11):1723-1732. doi: 10.1007/s00134-016-4447-8. Epub 2016 Sep 30. PMID 27686347